CLINICAL TRIAL: NCT03445260
Title: PeRioperative Optimization With Nutritional Supplements in Patients Undergoing GastRointEStinal Surgery for Cancer (PROGRESS): A Randomized Placebo Controlled Feasibility Study.
Brief Title: PeRioperative Optimization With Nutritional Supplements for Patients Undergoing GastRointEStinal Surgery for Cancer
Acronym: PROGRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Pablo Serrano, Assistant Professor, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3988
Record Dates: First submitted 2017-12-21; First posted 2018-02-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Each placebo is composed of a collagen-based filler with exactly the same taste and texture as the intervention.
  Interventions: Other: Placebo
- Nutritional Supplements (Experimental): carbohydrate loading, immunonutrition (formulated liquid diet), protein supplement
  Interventions: Other: Nutritional Supplements

INTERVENTIONS:
Other: Nutritional Supplements — PreCovery is a carbohydrate loading nutritional supplement, INergy FLD is an immunonutrition formulated liquid diet, and ISOlution is a protein supplement.
  Other Names: PreCovery; INergy FLD; ISOlution
  Arms: Nutritional Supplements
Other: Placebo — Each placebo is composed of a collagen-based filler with exactly the same taste and texture as the intervention.
  Arms: Placebo

SUMMARY:
This is a single-center randomized, placebo-controlled, double-blind feasibility study comparing the intervention of perioperative nutritional supplements (immunomodulation, carbohydrate loading, and protein isolate) with an identical placebo for each solution in patients with gastrointestinal cancer undergoing surgery. Eligible and consenting patients will be randomly allocated to receive the intervention or placebo in a 1:1 ratio.

This study will assess the feasibility of a large, multi-centre trial by establishing the feasibility of randomization to intervention or placebo. This study will be conducted at the Juravinski Hospital and will enroll 100 patients over 18 months.

The study intervention includes three perioperative nutritional supplements: (1) a protein supplement administered 3 times a day for 30 days before surgery, (2) a sugar-based supplement administered the day prior to and the day of surgery, and (3) a formulated liquid diet containing arginine, RNA, proteins and omega-6 fatty acids (referred to as immunonutrition for the purposes of this study) administered for 5 days prior to and 5 days after surgery.

The primary outcome for each eligible patient is defined as being randomized to intervention or placebo. The criteria for success of this study is defined as the proportion of eligible patients randomized as ≥ 60%. If the estimated proportion is <40%, the trial will be considered not feasible. If the proportion is between 40%-59%, the trial will be considered feasible with modifications to improve enrolment. Other secondary objectives include compliance with study intervention, estimating differences in postoperative complications, length of hospital stay, and quality of life between groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older
* Diagnosed with a resectable type of gastrointestinal cancer (e.g. cancers of the gallbladder, liver, pancreas, stomach, small intestine, colon and rectum) for which an elective operation is planned (resection vs. palliative procedure).
* Patients with distant metastasis are eligible for the study.
* Patients who are lactose intolerant are also eligible for the study because the amount of lactose in ISOlution and PreCovery is minimal (trace).

Exclusion Criteria:

* Malabsorption syndrome (e.g. chronic pancreatitis)
* Cannot tolerate oral intake (e.g. gastric outlet obstruction or delayed gastric emptying)
* Organ failure (liver, kidney); end stage liver disease with a Child Pugh Score ≥ B or end stage renal disease defined as stages 3 and 4 with a glomerular filtration rate between 30-59 for stage 3 and 15-29 for stage 4.
* Inflammatory diseases such as rheumatoid arthritis, systemic lupus erythematous, Crohn's disease and ulcerative colitis
* Patients currently on steroids
* Poorly controlled type 1 or 2 diabetes mellitus
* Female patients who are pregnant and/or lactating
* Galactosemia
* Ongoing infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The number of patients randomized to the study | 21 months
  Feasibility of this study will be determined by the number of eligible patients randomized to intervention or placebo.

SECONDARY OUTCOMES:
The number of patients who comply with the study intervention regimen | 30 days before index surgery, and up to 5 days after index surgery
  Compliance will be defined as intake of at least 70% of study intervention regimen.
Overall Complications | 3 months after index surgery
  Occurrence of any postoperative complication (major or minor) from surgery following each patient's hospital stay and up to 90 days from the initial operation. Occurrence of any postoperative infections will also be calculated.
Comprehensive Complication Index | 3 months after index surgery
  At 90 days from the index operation will be determined for each patient. This index can be calculated for each patient using the online calculator www.assessurgery.com25 following the grading of each postoperative complication according to Clavien-Dindo.
Quality of Life (QoL) - EORTC-QLQ-C Instrument | Baseline, 1 month, and 3 months after index surgery
  The global health related QoL at baseline, 1 and 3 months following randomization measured using the EORTC-QLQ-C instrument.
Quality of Life (QoL) - FACT-G Scale | Baseline, 1 month, and 3 months after index surgery
  The global health related QoL at baseline, 1 and 3 months following randomization measured using the FACT-G scale.
Length of Hospital Stay | 1 month after index surgery
  Will be determined for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serrano PE, Parpia S, Nair S, Ruo L, Simunovic M, Levine O, Duceppe E, Rodrigues C. Perioperative Optimization With Nutritional Supplements in Patients Undergoing Gastrointestinal Surgery for Cancer (PROGRESS): Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 31;7(10):e10491. doi: 10.2196/10491. PMID 30381282